CLINICAL TRIAL: NCT05432349
Title: Rett Syndrome Real World Data Observational Registry
Brief Title: Rett Syndrome Registry
Acronym: RSR
Status: Recruiting | Type: Observational
Sponsor: International Rett Syndrome Foundation (Other)
Collaborators: Boston Children's Hospital (Other); Children's Health UTSW (Unknown); Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other); Gillette Children's Specialty Healthcare (Other); Greenwood Genetic Center (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); Montefiore Medical Center (Other); Rush University (Other); St. Louis Children's Hospital (Other); Baylor College of Medicine (Other); University of Alabama at Birmingham (Other); UCSF Benioff Children's Hospital Oakland (Other); Vanderbilt University Medical Center (Other); Hive Networks (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00060206
Record Dates: First submitted 2022-04-05; First posted 2022-06-27 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Rett Syndrome; Rett Syndrome, Atypical; Genetic Disease; Genetic Diseases, X-Linked; Intellectual Disability; Neurobehavioral Manifestations; Neurologic Manifestations; Neurologic Disorder; Neurodevelopmental Disorders; Nervous System Diseases
Keywords: Rett syndrome; MECP2; Neurodevelopmental disorder; Registry; Natural History Study
MeSH Terms: conditions — Rett Syndrome; Rett Syndrome, Atypical; Genetic Diseases, Inborn; Genetic Diseases, X-Linked; Intellectual Disability; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Rett Syndrome Registry is a longitudinal observational study of individuals with MECP2 mutations and a diagnosis of Rett syndrome. Designed together with the IRSF Rett Syndrome Center of Excellence Network medical directors, this study collects data on the signs and symptoms of Rett syndrome as reported by the Rett syndrome experts and by the caregivers of individuals with Rett syndrome. This study will be used to develop consensus based guidelines for the care of your loved ones with Rett syndrome and to facilitate the development of better clinical trials and other aspects of the drug development path for Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a pathologic loss of function alteration of MECP2

Exclusion Criteria:

* Male or female with a gain of function alteration of MECP2, including those with MEPC2 duplication or triplication

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is males and females of all ages with a loss of function alteration of the MECP2 gene, most commonly resulting in Rett syndrome.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Natural History | 5 years
  To longitudinally evaluate the natural history of patients with mutations on the MECP2 gene, estimating and defining their clinical spectrum (e.g. disease course and complications of disease).

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, Oakland, California
  - Children's Hospital Colorado, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - The Children's Hospital at Montefiore, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt Kennedy Center, Nashville, Tennessee
  - Children's Health, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas